CLINICAL TRIAL: NCT02597816
Title: Three Dimensional Trans-vaginal Ultrasound to Reevaluate Arcuate Uteri Diagnosed by Hystro-salpingography
Brief Title: Role of Three Dimensional Ultrasound in the Diagnosis of Septate Uterus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohammed Khairy Ali, Dr, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TDU
Record Dates: First submitted 2015-11-04; First posted 2015-11-05 (Estimated); Last update posted 2015-12-18 (Estimated); Status verified 2013-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Three dimensional ultrasound (Other): Infertile women with diagnosis of arcuate and septate uterus based on Hystro-salpingography were recruited. All women were examined by Three dimensional ultrasound on day 22 cycle to allow for better delineation of the uterine contour. The outer and inner fundal contours and the length of the fundal notch were examined by Three dimensional ultrasound in the mid-coronal view of the multi-planar and multi-slice display of the uterus. The final diagnosis of the anomalies was based on combined hysteroscopy/laparoscopy examination, the gold standard.
  Interventions: Radiation: Three dimensional ultrasound

INTERVENTIONS:
Radiation: Three dimensional ultrasound

SUMMARY:
Congenital uterine anomalies are found in 8% of infertile women and 24.5% of infertile women with a history of recurrent miscarriage, with septate and sub-septate uterus being the most common anomalies in these women, Also, septate uterus is the commonest anomaly found in infertile women requiring assisted reproductive technology.

Published data showed improved Cumulative pregnancy rate and live birth rate, and a significant reduction in Miscarriage rate in In Vitro Fertilization women after hysteroscopic metroplasty of both small and large septate compared to non-operated women.

Investigators hypothesized that trans-vaginal three Dimensional Ultrasound will be superior to Hystro-salpingography for the differentiation between arcuate and septate uterus in infertile women scheduled for In Vitro Fertilization.

ELIGIBILITY:
Inclusion Criteria:

* women with primary infertility,
* an indication for IVF and
* Suspected arcuate or septate uterus diagnosis based on hysterosalpingography .

Exclusion Criteria:

* were confirmed uterine abnormality by prior office hysteroscopy

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2013-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Number of patients diagnosed to have subseptate uterus by three dimensional ultrasound | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut university, Asyut, Egypt